CLINICAL TRIAL: NCT02336620
Title: Balanced Salt Solution Versus Normal Saline Solution During Initial Resuscitation in Severe Sepsis or Septic Shock Children: A Randomized Controlled Trial
Brief Title: Balanced Salt Solution VS. Normal Saline Solution in Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Nattachai Anantasit, Pediatric Department, Ramathibodi Hospital, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RF_58015
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Shock, Septic; Sepsis
Keywords: Severe sepsis, Balanced Salt Solution, Normal Saline
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ringer Acetate (Experimental): Ringer acetate 10-20 ml/kg IV bolus when patient need fluid bolus
  Interventions: Drug: Ringer acetate
- Normal saline (Active Comparator): NSS 10-20 ml/kg IV bolus when patient need fluid bolus
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ringer acetate — Ringer acetate 10-20 ml/kg IV bolus in 15-30 min,repeat bolus as needed by patient status
  Arms: Ringer Acetate
Drug: Normal saline — NSS 10-20 ml/kg IV bolus in 15-30 min,repeat bolus as needed by patient status
  Other Names: NSS
  Arms: Normal saline

SUMMARY:
The Purpose of this study is to determine the impact of balanced salt solution versus chloride rich solution on clinical outcomes in paediatric severe sepsis or septic shock

DETAILED DESCRIPTION:
The surviving sepsis campaign guideline recommended the isotonic crystalloids as the first choice of initial fluid resuscitation. The isotonic crystalloids are including chloride-rich solution (eg.NSS) and balanced salt solution. Retrospective study showed normal saline can induced hyperchloremic metabolic acidosis and acute kidney injury. However, no randomized controlled trial compare efficacy between the balanced salt solution and chloride rich solution.

ELIGIBILITY:
Inclusion Criteria:

* children younger than 18 year old who has severe sepsis or septic shock
* inform consent

Exclusion Criteria:

* children who had shock from other aetiologies
* end stage disease or severe congenital anomaly
* refuse to inform consent

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
incidence of hyperchloremic metabolic acidosis | 48 hour

SECONDARY OUTCOMES:
28 day and 90 day mortality rate | 28 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Anantasit, M.D., Principal Investigator — Ramathibodi Hospital, Bangkok
Locations (1):
- Department of Pediatric,Ramathibodi Hospital, Bangkok, Thailand